CLINICAL TRIAL: NCT06848088
Title: Extended Follow-up of Patients With Melanoma Treated With Fianlimab Plus Cemiplimab in Expansion Cohorts From Study R3767-ONC-1613
Brief Title: A Study to Learn About the Long-Term Health of Adult Participants From a Previous Study of a New Melanoma Treatment
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R3767-ONC-2466; 2024-517729-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
Keywords: Advanced Skin Cancer
MeSH Terms: conditions — Melanoma | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- With Disease Progression at Enrollment (Other)
  Interventions: Drug: Fianlimab+cemiplimab
- No Progressive Disease at Enrollment (Other)
  Interventions: Drug: Fianlimab+cemiplimab

INTERVENTIONS:
Drug: Fianlimab+cemiplimab — No study drug administered in this observational study.
  Other Names: REGN3767; REGN2810; Libtayo®

SUMMARY:
This study is researching the long-term effects of a combination of experimental drugs called fianlimab and cemiplimab. The study is being conducted in patients with advanced skin cancer (melanoma) who had previously been treated with fianlimab and cemiplimab in the study called R3767-ONC-1613 (NCT03005782).

The aim of the current study is to see how safe and effective the study drugs are in a long-term follow-up. No study drug will be given during this study. Cancer status will be monitored, in addition to routine care. The study is also collecting information about general health status, and other treatments that may have been received since participation in study R3767-ONC-1613 (NCT03005782).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with melanoma who enrolled in cohorts 6, 15, or 16 of study R3767-ONC- 1613 (NCT03005782)

Key Exclusion Criteria:

None

Note: Other protocol-defined Inclusion/ Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2029-10-10 (Estimated); Study Completion 2029-10-10 (Estimated)

PRIMARY OUTCOMES:
Death from any cause starting at time of initial treatment with fianlimab and cemiplimab in study R3767-ONC-1613 | Up to 4 years

SECONDARY OUTCOMES:
Progressive-Free Survival (PFS) | Up to 4 years
Objective Response Rate (ORR) | Up to 4 years
Duration of Response (DOR) | Up to 4 years
Disease Control Rate (DCR) | Up to 4 years
Incidence of Serious Adverse Events (SAEs) | Up to 4 years
Severity of SAEs | Up to 4 years
Incidence of treatment-related AEs | Up to 4 years
Severity of treatment-related AEs | Up to 4 years
Incidence of anti-cancer therapies received since end of treatment with fianlimab and cemiplimab in study R3767-ONC-1613 | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (8):
- United States (7):
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Oncology And Hematology, San Antonio, Texas
- St. Vincent's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/